CLINICAL TRIAL: NCT05768867
Title: French Translation and Validation of the PEYronie's Disease QUESTionnaire
Acronym: FRAPEYQUEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0012; 2023-A00219-36 (Registry Identifier: ANSM)
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Peyronie Disease
MeSH Terms: conditions — Penile Induration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: FRAnçaise du PEYronie's Disease QUESTionnaire — Complete an online FRAnçaise du PEYronie's Disease QUESTionnaire

SUMMARY:
This study is a prospective cohort dedicated to peyronie's disease. The aim is to validate the french translation of the peyronie's disease questionnaire. The primary endpoint is the response rate to the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient with Peyronie's Disease clinically diagnosed during a consultation, with palpation of at least one plaque

Exclusion Criteria:

* Patient refusing to participate
* Patient with difficulties in understanding the French language.
* Protected persons referred to in articles L.1121-6 to L.1121-8 of the public health code

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Peyronie's Disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Rate of responses | Day 0
  Response rate to the online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Huyghe, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Toulouse Hospital, Toulouse, France